CLINICAL TRIAL: NCT01364740
Title: PMP-300E: Validation of Portable Monitoring Device PMP-300E for Identification of Obstructive Sleep Apnea.
Brief Title: PMP-300E (Smart Watch): Portable Monitoring Device Study
Acronym: PMP-300E
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Clete A. Kushida, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-04212009-2358; K073327 (Registry Identifier: clinicaltrials.stanford.edu); SPO 42154 (Other: Stanford University, OSR); eProtocol 13181 (Other: Stanford University, IRB)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PMP-300E, In-Lab PSG (Experimental): PMP-300E, A 7-channel (nasal pressure, effort, snoring, SpO2, pulse rate, body position and movement) Level 3 portable monitor (11.2 x 3.3 x 5.5cm, 80g, Pacific Medico Co., LTD) to measure sleep-related breathing will be tested against conventional gold-standard In-Lab Polysomnography (sleep study)
  Interventions: Device: PMP-300E; Device: In-lab PSG

INTERVENTIONS:
Device: PMP-300E — Data collected from Level 3 device
  Other Names: SmartWatch; Portable Monitoring Device; Sleep Apnea; Home Study; Sleep Diagnostic Device
Device: In-lab PSG — Data collected from Type I In-Lab Polysomnography
  Other Names: Sleep Study

SUMMARY:
Validation of Portable Monitoring Device PMP-300E for Identification of Obstructive Sleep Apnea.

DETAILED DESCRIPTION:
The purpose of the study is to validate an Obstructive Sleep Apnea portable monitoring device, PMP-300E. Validating process compared data collected by PMP-300E with data collected from in-lab polysomnography.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Age 18 and over.
* Require a sleep diagnostic study by physician's order.
* Able and willing to provide written informed consent.
* Able to speak and read English.

Exclusion Criteria:Exclusion Criteria:

* Participation in another interventional research study within the last 30 days.
* Unstable medical or psychiatric conditions that would interfere with the demands of the study or the ability to commit to follow-up assessment. Examples include unstable congestive heart failure, neuromuscular disease, cancer, and renal failure.
* Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate or severe COPD or other pulmonary disorders, or any condition with an elevation of arterial carbon dioxide levels (> 45 mmHg) while awake or participants qualifying for oxygen therapy (arterial saturation 88% for more than five minutes).
* Consumption of ethanol more than 4 nights per week. (CAGE criteria)
* Use of recreational drug within the past 12 months.
* Women who are pregnant or currently lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clete A. Kushida M.D., Ph.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Center for Human Sleep Research, Redwood City, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through the patient population at the Stanford Sleep Medicine Center
Groups:
- SmartWatch PMP-300E: Investigational device Smart Watch PMP-300E to measure sleep-related breathing was tested against conventional gold-standard In-Lab Polysomnography (sleep studies)
  Smart Watch PMP-300E: Data collected from a Level 3 portable monitoring device
  In-lab Polysomnography: Data collected from Type I In-Lab Polysomnography
Period: Overall Study
Arm/Group | SmartWatch PMP-300E
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PMP-300E, In-Lab PSG: PMP-300E, In-Lab PSG: PMP-300E, A 7-channel (nasal pressure, effort, snoring, SpO2, pulse rate, body position and movement) Level 3 portable monitor (11.2 x 3.3 x 5.5cm, 80g, Pacific Medico Co., LTD) to measure sleep-related breathing will be tested against conventional gold-standard In-Lab Polysomnography (sleep study)
  PMP-300E: Data collected from Level 3 device
  In-lab PSG: Data collected from Type I In-Lab Polysomnography
Arm/Group | PMP-300E, In-Lab PSG
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years]
  Men | 54.3 (15.46)
  Women | 56.8 (14.24)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2]
  Men | 29.5 (9.54)
  Women | 30.8 (11.76)
Epworth Sleepiness Scale score [Mean (Standard Deviation); unit: units on a scale] — Subjective measure of daytime sleepiness, 0-24 points, where higher numbers indicate greater levels of subjective daytime sleepiness
  units on a scale | 6.9 (5.61)

OUTCOME MEASURES:

1. Primary Outcome: AHI
Description: Apnea-Hypopnea Index (number of events/hour of sleep). Hypopneas scored without EEG arousals.
Time Frame: One night
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- PMP-300E, In-Lab Polysomnography: Patient data from one night with the PMP-300E, compared to In-Lab PSG data
Arm/Group | PMP-300E, In-Lab Polysomnography
Number analyzed (Participants) | 10
events/hour
  PMP-300E | 19.2 (14.50)
  In-Lab PSG | 19.3 (14.5)
Statistical Analysis 1: Comparison: PMP-300E, In-Lab Polysomnography; Patient data from one night with the PMP-300E compared to In-Lab PSG data; Test type: Superiority or Other; p > 0.05, Sign test

2. Secondary Outcome: Apnea Index
Description: Number of events/hour of sleep
Time Frame: One night
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | PMP-300E, In-Lab Polysomnography
Number analyzed (Participants) | 10
events/hour
  PMP-300E | 7.7 (11.06)
  In-Lab PSG | 9.8 (13.32)
Statistical Analysis 1: Comparison: PMP-300E, In-Lab Polysomnography; Patient data from one night with the PMP-300E compared to In-Lab PSG data; Test type: Superiority or Other; p > 0.05, Sign test

3. Secondary Outcome: Hypopnea Index
Description: Number of events/hour of sleep. Hypopneas scored without EEG arousals.
Time Frame: One night
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | PMP-300E, In-Lab Polysomnography
Number analyzed (Participants) | 10
events/hour
  PMP-300E | 8.8 (4.96)
  In-Lab PSG | 14.1 (19.0)
Statistical Analysis 1: Comparison: PMP-300E, In-Lab Polysomnography; Patient data from one night with the PMP-300E compared to In-Lab PSG data; Test type: Superiority or Other; p > 0.05, Sign test

4. Secondary Outcome: Oxygen Saturation
Description: Mean oxygen saturation
Time Frame: One night
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | PMP-300E, In-Lab Polysomnography
Number analyzed (Participants) | 10
percent
  PMP-300E | 94.8 (2.10)
  In-Lab PSG | 95.0 (2.11)
Statistical Analysis 1: Comparison: PMP-300E, In-Lab Polysomnography; Patient data from one night with the PMP-300E compared to In-Lab PSG data; Test type: Superiority or Other; p > 0.05, Sign test

5. Other Pre Specified Outcome: Attitude Toward Device Use Questionnaire Scores
Description: Questionnaire consisting of multiple questions, scored as 1 = disagree completely to 5 = agree completely, revealed the following mean scores
Time Frame: one night
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- PMP-300E: Patient questionnaire data collected after one night with the PMP-300E
Arm/Group | PMP-300E
Number analyzed (Participants) | 10
units on a scale
  Confident in using device at home | 4.3 (0.82)
  Confident in applying nasal cannula on own | 4.4 (0.84)
  confident in applying finger probe on own | 4.9 (0.32)
  Can read window display without difficulty | 3.9 (0.99)
  Can hear the on/off beep without difficulty | 3.8 (1.03)
  Can strap on chest belt without difficulty | 4.5 (0.71)
  Importance of finding out more about own sleep | 4.8 (0.42)
  Bed partner is a restless sleeper or loud snorer | 1.2 (1.40)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | PMP-300E, In-Lab Polysomnography
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No